CLINICAL TRIAL: NCT02430558
Title: Second Line Treatment of Knee Osteochondral Lesion With Decellularized Treated Osteochondral Allograft. Phase IIa Trial
Brief Title: Second Line Treatment of Knee Osteochondral Lesion With Treated Osteochondral Graft
Acronym: ODPHOENIX2
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low accrual rate
Sponsor: TBF Genie Tissulaire (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-A00002-47
Record Dates: First submitted 2015-04-25; First posted 2015-04-30 (Estimated); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Cartilage Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OD-PHOENIX (Experimental): treatment of 1 to 5 osteochondral allograft cylinders in mosaic
  Interventions: Biological: OD-PHOENIX

INTERVENTIONS:
Biological: OD-PHOENIX — Decellularized, freeze-dried, irradiated osteochondral allograft
  Other Names: Osteochondral allograft

SUMMARY:
Patient with IKDC score < 65, pretreated with mosaicplasty or ACI ( with matrix or not) within > 18 months, with one or two osteochondral lesions are recruited to have treated osteochondral allografts in mosaicplasty.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between the ages of 18 and 55

  * osteochondral lesions of the knee due to trauma or osteochondritis dissecans or removal treatment ( lesion post autograft)
  * Osteochondral lesion > grade II- ICRS
  * One lesion or 2 concomitant lesions (tibial plateau, patella and condyles )at least one lesion has been pretreated by mosaicplasy or ACI. These treatment would have to have been made at least 18 months before inclusion
  * Presence of disabling and clinically meaningful symptoms (subjective IKDC < 65, no improvement for 3 months)
  * No significant obesity (BMI < 30)
  * Accompanying ligamentous and meniscal lesions, joint malalignment and patella femoral instability are authorized and corrected concurrently.
  * Patient able to understand, sign and date the informed consent form
  * Patient affiliated with a national health insurance system or who is the beneficiary of such as system
  * Women of childbearing age may not be included in the clinical trial unless their pregnancy test is negative. If this test is negative, they will be asked to use an effective birth control method during the entire the study.

Exclusion Criteria:

* - Pregnant or breast feeding women: Women of childbearing age will be asked to undergo a pregnancy test before being enrolled into the study and to use an effective birth control method.
* Presence of osteoarthritis, rheumatoid arthritis, any other condition of knee joint that, in the surgeon's opinion, is likely to compromise the allograft's outcome
* Excessive laxity or recurrent instability that could affect the score evaluation without concomitant ligamentoplasty
* Presence of an ulcerative disease, heavy smoking, tuberculosis, chronic psychiatric disorder or disease requiring long-term treatment with a medication that would affect bone or joint metabolism
* Persons with cancer or a history of cancer
* Persons deprived of their freedom by a judicial or administrative decision
* Adults subject to legal protection measures or who are unable to provide their consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-04-05 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
improvement of IKDC score | 18 months

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 18 months
recellularization of tissue (arthroscopy and histology) | 18 months
  arthroscopy and histology
integration of the tissue by imagery | 18 months